CLINICAL TRIAL: NCT01349101
Title: Post Transplant Cyclophosphamide for Unrelated and Related Allogeneic Hematopoietic Stem Cell Transplantation for Hematological Malignancies
Brief Title: A Research Study of Bone Marrow Transplantation From Unrelated or Partially Matched Related Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11D.51; 2010-54 (Other: CCRRC); JT 2137 (Other: JeffTrial Number)
Record Dates: First submitted 2011-04-26; First posted 2011-05-06 (Estimated); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Hematological Malignancies
Keywords: hematopoietic stem cell transplantation; HSCT; allogeneic marrow transplantation; cyclophosphamide; graft-versus-host disease; GVHD
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease | interventions — Whole-Body Irradiation; Radiotherapy; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; fludarabine; fludarabine phosphate; Busulfan; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myeloablative HSCT (Experimental): Myeloablative Hematopoietic Stem Cell Transplantation (HSCT): Patients will receive myeloablative transplants or nonmyeloablative transplants depending on their disease type.
  Interventions: Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Genetic: Hematopoietic stem cell transplantation
- Reduced Intensity HSCT (Experimental): Reduced Intensity Hematopoietic Stem Cell Transplantation (HSCT): Patients who have received a previous transplant, patients who have received dose limiting radiation, and patients with a DLCO <45% will receive the reduced intensity conditioning regimen.
  Interventions: Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Fludarabine; Drug: Busulfan; Genetic: Hematopoietic stem cell transplantation

INTERVENTIONS:
Radiation: Total Body Irradiation — Myeloablative HSCT Arm: Total body irradiation (TBI) is given in 8 fractions over 4 days (total dose of 12 Gy)
  Reduced Intensity HSCT Arm: TBI is given in one fraction (total dose of 2 Gy)
  Other Names: TBI; radiotherapy
Drug: Cyclophosphamide — Cyclophosphamide is administered on the third day after the hematopoietic stem cell transplantation (HSCT) to help reduce graft-versus-host disease (GVHD). It is given at a dose of 60 mg/kg/d for 2 days on days +3 and +4.
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; Cytophosphane; Cy
Drug: Tacrolimus — Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Other Names: FK-506; Fujimycin
Drug: Mycophenolate mofetil — Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Other Names: CellCept; MMF
Drug: Fludarabine — Started the fifth day before the transplant. Given for four days at 30 mg/m2/d.
  Other Names: fludarabine phosphate; Fludara
  Arms: Reduced Intensity HSCT
Drug: Busulfan — Started the fourth day before the transplant. Given for two days at 3.2 mg/kg.
  Other Names: Myleran, Busulfex IV
  Arms: Reduced Intensity HSCT
Genetic: Hematopoietic stem cell transplantation — Allogeneic marrow transplantation given after the last dose of total body irradiation (TBI)
  Other Names: HSCT

SUMMARY:
It is hypothesized that engraftment when administering cyclophosphamide post the stem cell infusion will increase, the incidence of graft versus host disease (GVHD) and day 100 mortality will decrease, and the use of cyclophosphamide post stem cell infusion with alternative donors will be as safe and as effective as traditional matched transplants.

DETAILED DESCRIPTION:
The primary rationale for the development of this research study is to find out if the use of cyclophosphamide after a "blood" stem cell transplant is an effective treatment for patients with blood cancers who require transplant for long-term survival but are without an available matched-sibling donor. Historically, survival rates for patients undergoing partially matched related or unrelated donor transplants (henceforth to be called alternative donor transplants) have been much lower than those observed after matched sibling stem cell transplants. Survival post alternative donor stem cell transplant has also been affected by the requirement to remove or reduce the numbers of donor T cells resulting in higher rates of infection, graft rejection, and relapse. One significant limitation to conventional donor transplants with HLA matched siblings has been that over 50% of patients do not have HLA matched siblings so that increasing the safety of alternative donor transplants could have a significant influence on the number of patients who could safely receive transplants. Because of the historically low overall survival (OS) after alternative donor transplants, it has become a procedure of "last resort" in many centers unwilling to consider it unless all other options are exhausted. There fore several centers including ours have sought to overcome problems using various strategies. The strategy the investigators have proposed for this study (which has been used similarly by other centers) has been to administer cyclophosphamide post the stem cell infusion (traditionally it is given before the stem cell infusion) thereby hopefully destroying the activated T-cells causing graft-versus host disease (GVHD) and allow T cell tolerization and engraftment; but, not the inactivated T cells thereby hopefully preserving the anti-tumor effects of the donor immune system. Thus, the major aim of this study will be to measure the engraftment with this regimen and secondarily to measure incidence of GVHD and day 100 mortality. The goal is to see if in the first 3 months the use of cyclophosphamide post stem cell infusion with alternative donors is as safe and as effective as traditional matched transplants.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a hematological or oncological diagnosis in which allogeneic hematopoietic stem cell transplantation (HSCT) is thought to be beneficial.

   1. Patients without morphological or molecular evidence of disease
   2. For patients with "indolent diseases," if the patient has evidence of disease the disease burden must be minimal (at least PR) and the disease must be chemoresponsive. Thus for example patients with acute leukemia (not an indolent disease) must be in a morphological CR or CRp.
2. For patients with MDS the inclusion criteria is specifically as follows:

   * For patients with RA or RARS or isolated 5q- they can proceed to transplant without any treatment.
   * For patients with RAEB-1, RCMD+/-RS, or MDS NOS must have stable disease for 6 months (as documented by serial bone marrow examinations) in the absence of any therapy but growth factors or transfusion support. Patients who require treatment to "control their disease" must show chemo-responsiveness
   * For patients with CMML or RAEB-2 they must demonstrate chemo-responsiveness
   * Chemo-responsiveness is defined as a blast percentage decrease by at least 5 percentage points and there must be less than 10% blasts after treatment and at the time of transplant, if there are more than 10% blasts at any point during the disease course
   * Chemo-responsiveness must also include at least one of the following if applicable:

     * A cytogenetic response
     * A well-documented decrease in transfusion requirements.
3. Patients must have a related donor who is zero, one, two, three, or four antigen mismatched at the HLA-A; B; C; DR loci or an unrelated donor up to a two antigen mismatch. DNA will be retained by the tissue typing laboratory for possible typing for DQ and DP. When multiple related donor options are available donor selection will be determined the same as in the TJU two-step protocols. When multiple unrelated donors are available care will be made to avoid HLA-A and HLA-B mismatches if possible based on data from the Japanese Marrow Donor Registry studies. An HLA antibody screen will be performed on each patient.
4. All patients must have adequate organ function:

   1. Patients with related donors must have an LVEF of >35%. Patients with unrelated donors must have an LVEF >45%. Patients with LVEF ≤50% and all patients with symptoms or history of heart failure or coronary artery disease must have a stress echo or equivalent test and a cardiological evaluation.
   2. Patients with related donors must have a DLCO >35% of predicted corrected for hemoglobin. Patients with unrelated donors must have a DLCO >45% of predicted corrected for hemoglobin. For related donors if the DLCO is less than 45% the EF must be greater than 45% and vice versa.
   3. Patients with related donors must have an adequate liver function as defined by a serum bilirubin <3.0, AST and ALT <3.0X upper limit of normal. Patients with unrelated donors must have an adequate liver function as defined by a serum bilirubin <1.8, AST and ALT < 2.5X upper limit of normal. Exceptions may be granted for patients with "benign" liver disorders such as Gilbert's disease.
   4. Patients with related donors or with unrelated donors must have a creatinine clearance of > 60 ml/min/1.73 m^2.
   5. Patients with related donors must have a performance status > 60% (TJU Karnofsky14) (Appendix A). Patients with unrelated donors must have a Performance status > 70% (TJU Karnofsky).
   6. Patients with related donors must have a HCT-CI Score < 6 Points (Appendix B). Patients with unrelated donors must have a HCT-CI Score < 5 Points.
   7. Patients must be willing to use contraception if they are of childbearing potential.
   8. Patients must be able to give informed consent or have a care giver who can give consent.
   9. Patients that are HIV positive will be eligible for the study if they have an undetectable viral load and meet the above criteria for patients with unrelated donors.

Exclusion Criteria:

1. Patients with related donors who have a combination of Performance status of < 70% (TJU Karnofsky) and an HCT-CI of 4 points or more. Patients with unrelated donors with a combination of Performance status of < 80% (TJU Karnofsky) and an HCT-CI of 4 points or more.
2. Patients with active involvement of the central nervous system with malignancy. Patients with a disease with potential for CNS involvement should have documentation of the lack of CNS involvement via lumbar puncture or similar procedure performed within two months of admission or as per TJU standard practice guidelines.
3. Patients with a psychiatric disorder that would preclude patients from complying with the protocol even with a caregiver. Patients with a lack of social support that would interfere with the ability to receive appropriate medical care will also be excluded.
4. Pregnancy
5. Patients with life expectancy of < 6 months for reasons other than their underlying hematological/oncological disorder.
6. Patients who have received alemtuzumab within 8 weeks of the transplant admission, or who have recently received horse or rabbit ant-thymocyte globulin and have an ATG level of > 2 μg/ml. Patients on systemic corticosteroids at a dose equivalent of prednisone 7.5mg/day or higher.
7. Patients who cannot receive cyclophosphamide.
8. Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol.
9. Patients with refractory disease.
10. Patients with clinically significant preformed antibodies to their donors.
11. Patients who require supplemental oxygen other than for sleep apnea will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-02-10 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L Wagner, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Myeloablative HSCT: Myeloablative Hematopoietic Stem Cell Transplantation (HSCT): Patients will receive myeloablative transplants or nonmyeloablative transplants depending on their disease type.
  Total Body Irradiation: Myeloablative HSCT Arm: Total body irradiation (TBI) is given in 8 fractions over 4 days (total dose of 12 Gy)
  Cyclophosphamide: Cyclophosphamide is administered on the third day after the hematopoietic stem cell transplantation (HSCT) to help reduce graft-versus-host disease (GVHD). It is given at a dose of 60 mg/kg/d for 2 days on days +3 and +4.
  Tacrolimus: Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Mycophenolate mofetil: Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Hematopoietic stem cell transplantation: Allogeneic marrow transplantation given after the last dose of total body irradiation (TBI)
- Reduced Intensity HSCT: Reduced Intensity Hematopoietic Stem Cell Transplantation (HSCT): Patients who have received a previous transplant, patients who have received dose limiting radiation, and patients with a DLCO <45% will receive the reduced intensity conditioning regimen.
  Total Body Irradiation: Reduced Intensity HSCT Arm: TBI is given in one fraction (total dose of 2 Gy)
  Cyclophosphamide: Cyclophosphamide is administered on the third day after the hematopoietic stem cell transplantation (HSCT) to help reduce graft-versus-host disease (GVHD). It is given at a dose of 60 mg/kg/d for 2 days on days +3 and +4.
  Tacrolimus: Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Mycophenolate mofetil: Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Fludarabine: Started the fifth day before the transplant. Given for four days at 30 mg/m2/d.
  Busulfan: Started the fourth day before the transplant. Given for two days at 3.2 mg/kg.
  Hematopoietic stem cell transplantation: Allogeneic marrow transplantation given after the last dose of total body irradiation (TBI)
Period: Overall Study
Arm/Group | Myeloablative HSCT | Reduced Intensity HSCT
Started | 33 | 45
Completed | 29 | 36
Not Completed | 4 | 9
Not completed — Disease Progression | 1 | 1
Not completed — Death | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myeloablative HSCT | Reduced Intensity HSCT | Total
Number analyzed (Participants) | 33 | 45 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 17 | 50
  >=65 years | 0 | 28 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 16 | 24 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 28 | 44 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 21 | 38 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Successful Engraftment Using Cyclophosphamide Post-Transplant
Description: Successful Hematopoietic engraftment will be assessed by determining the incidence of participants who achieve both of the following criteria within the 100 days post-transplant:
  ANC >/= 0.5x10e9/L for at least 3 days. Platelet engraftment >20,000 with no transfusions X 7 days. The incidence will be calculated as the number of participants who meet both engraftment criteria. Results will be presented as a proportion/percentage/probability not as an incidence rate.
Time Frame: Through 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: Cumulative Probability of Engraftment
Arm/Group | Myeloablative HSCT | Reduced Intensity HSCT
Number analyzed (Participants) | 33 | 45
Cumulative Probability of Engraftment | 1.00 [1.00 to 1.00] | 0.93 [0.86 to 1.00]

2. Secondary Outcome: Cumulative Incidence of Grade III-IV GVHD
Description: The cumulative incidence of Grade III-IV graft-versus-host disease (GVHD) within 100 days post-transplant will be estimated; goal is less than 10%. The cumulative incidence represents the probability that a participant experiences Grade III-IV GVHD by day 100. Results will be reported as proportion/percentage/probability.
Time Frame: Through 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: Cumulative Probability of Grade III-IV G
Arm/Group | Myeloablative HSCT | Reduced Intensity HSCT
Number analyzed (Participants) | 33 | 45
Cumulative Probability of Grade III-IV G | 0.5152 [0.3312 to 0.6716] | 0.3111 [0.1820 to 0.4493]

3. Secondary Outcome: Incidence of GVHD Unresponsive to Corticosteroids and Photopheresis
Description: This outcome will estimate the cumulative incidence (probability) of graft-versus-host disease (GVHD) that is considered unresponsive to corticosteroids and photopheresis within 100 days after treatment; goal is less than 15%. The cumulative incidence will be calculated as the number of participants meeting these criteria. Results will be reported as a proportion/percentage.
Time Frame: Through 100 days post-treatment
Measure: Number (95% Confidence Interval); unit: Cumulative Probability of GVHD
Arm/Group | Myeloablative HSCT | Reduced Intensity HSCT
Number analyzed (Participants) | 33 | 45
Cumulative Probability of GVHD | 0.0625 [0.0107 to 0.1838] | 0.0233 [0.00177 to 0.1072]

4. Secondary Outcome: Transplant-Related Mortality
Description: The cumulative incidence of transplant related mortality (TRM) by day 100 post-transplant will be estimated. Assess day 100 transplant-related mortality; goal is less than 15%. TRM is defined as death that results from medical treatment rather than from the underlying disease itself. The cumulative incidence reflects the probability of TRM by day 100. The result will be reported as a proportion/percentage/probability, not an incidence rate.
Time Frame: 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: Cumulative Probability of Mortality
Groups:
- Myeloablative HSCT: Myeloablative Hematopoietic Stem Cell Transplantation (HSCT): Patients will receive myeloablative transplants or nonmyeloablative transplants depending on their disease type.
  Total Body Irradiation: Myeloablative HSCT Arm: Total body irradiation (TBI) is given in 8 fractions over 4 days (total dose of 12 Gy)
  Reduced Intensity HSCT Arm: TBI is given in one fraction (total dose of 2 Gy)
  Cyclophosphamide: Cyclophosphamide is administered on the third day after the hematopoietic stem cell transplantation (HSCT) to help reduce graft-versus-host disease (GVHD). It is given at a dose of 60 mg/kg/d for 2 days on days +3 and +4.
  Tacrolimus: Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Mycophenolate mofetil: Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Hematopoietic stem cell transplantation: Allogeneic marrow transplantation given after the last dose of total body irradiation (TBI)
- Reduced Intensity HSCT: Reduced Intensity Hematopoietic Stem Cell Transplantation (HSCT): Patients who have received a previous transplant, patients who have received dose limiting radiation, and patients with a DLCO <45% will receive the reduced intensity conditioning regimen.
  Total Body Irradiation: Myeloablative HSCT Arm: Total body irradiation (TBI) is given in 8 fractions over 4 days (total dose of 12 Gy)
  Reduced Intensity HSCT Arm: TBI is given in one fraction (total dose of 2 Gy)
  Cyclophosphamide: Cyclophosphamide is administered on the third day after the hematopoietic stem cell transplantation (HSCT) to help reduce graft-versus-host disease (GVHD). It is given at a dose of 60 mg/kg/d for 2 days on days +3 and +4.
  Tacrolimus: Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Mycophenolate mofetil: Started the fifth day after the transplant to help prevent graft-versus-host disease (GVHD).
  Fludarabine: Started the fifth day before the transplant. Given for four days at 30 mg/m2/d.
  Busulfan: Started the fourth day before the transplant. Given for two days at 3.2 mg/kg.
  Hematopoietic stem cell transplantation: Allogeneic marrow transplantation given after the last dose of total body irradiation (TBI)
Arm/Group | Myeloablative HSCT | Reduced Intensity HSCT
Number analyzed (Participants) | 33 | 45
Cumulative Probability of Mortality | 0.0909 [0.0226 to 0.2192] | 0.1951 [0.0904 to 0.3292]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for 100 days following transplant.
Arm/Group | Myeloablative HSCT | Reduced Intensity HSCT
All-Cause Mortality (participants affected / at risk) | 3/33 | 8/45
Serious Adverse Events (participants affected / at risk) | 5/33 | 5/45
Other Adverse Events (participants affected / at risk) | 33/33 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative HSCT (N=33) | Reduced Intensity HSCT (N=45)
Acute Kidney Injury - Grade 3 (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute Kidney Injury - Grade 4 (Renal and urinary disorders) | 1 (1) | 5 (5)
Adenovirus - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
altered mental status - grade 4 (Psychiatric disorders) | 0 (0) | 1 (1)
Angioedema - Grade 4 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arterial Thrombosis - Grade 3 (Vascular disorders) | 0 (0) | 1 (1)
Atrial Fibrillation - Grade 2 (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation - Grade 3 (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete - grade 4 (Cardiac disorders) | 1 (1) | 0 (0)
BK Viremia - Grade 3 (Infections and infestations) | 1 (1) | 1 (1)
Blood bilirubin increased - Grade 3 (Hepatobiliary disorders) | 1 (1) | 0 (0)
Candidemia - Grade 3 (Infections and infestations) | 0 (0) | 1 (1)
Cardiomyopathy - Grade 3 (Cardiac disorders) | 1 (1) | 1 (1)
CMV Reactivation - Grade 4 (Infections and infestations) | 0 (0) | 1 (1)
CMV Viremia - Grade 3 (Infections and infestations) | 0 (0) | 1 (1)
Confusion - Grade 4 (Psychiatric disorders) | 1 (1) | 1 (1)
Creatinine increased - Grade 3 (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis - Grade 3 (Renal and urinary disorders) | 1 (1) | 0 (0)
Cytokine Release Syndrome - Grade 4 (Immune system disorders) | 0 (0) | 1 (1)
Decreased Ejection Fraction - Grade 3 (Cardiac disorders) | 1 (1) | 0 (0)
Delayed engraftment - Grade 3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Depressed Level of Consciousness - Grade 2 (General disorders) | 0 (0) | 1 (1)
Diarrhea -Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea - Grade 3 (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspnea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated Liver Function Tests - Grade 3 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Emesis - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Emesis - Grade 3 (Gastrointestinal disorders) | 1 (1) | 1 (1)
Failure to thrive - Grade 3 (General disorders) | 1 (1) | 0 (0)
Fatigue - Grade 3 (General disorders) | 1 (1) | 0 (0)
Fever - Grade 1 (Immune system disorders) | 0 (0) | 1 (1)
Fever - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Fever - Grade 3 (Immune system disorders) | 1 (1) | 0 (0)
Hypervolemia - Grade 3 (Vascular disorders) | 1 (1) | 0 (0)
Fungal Infection - Grade 4 (Infections and infestations) | 0 (0) | 1 (1)
Fungal PNA Nodules - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
Nausea - Grade 3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Graft rejection - Grade 4 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hearing impaired - Grade 2 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Heart failure - Grade 4 (Cardiac disorders) | 0 (0) | 1 (1)
Hematuria - Grade 3 (Renal and urinary disorders) | 1 (1) | 0 (0)
HHV-6 Infection - Grade 4 (Infections and infestations) | 1 (1) | 1 (1)
Singultus - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperbilirubinemia - Grade 3 (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperbilirubinemia - Grade 4 (Hepatobiliary disorders) | 1 (1) | 3 (4)
Hypervolemia - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Hypotension - Grade 2 (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension - Grade 4 (Cardiac disorders) | 1 (2) | 4 (4)
Hypoxia - Grade 2 (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypoxia - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Hypoxia - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4)
Increased Acute Rheumatic Fever - Grade 4 (Cardiac disorders) | 0 (0) | 1 (1)
increased creatinine - Grade 4 (Renal and urinary disorders) | 0 (0) | 3 (3)
Increased Liver Function Tests - Grade 4 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Infusion Related Reaction - chills - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - fever - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Hives - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - hypotension - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Hypoxia - Grade 3 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Pruritus - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - tachycardia - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Interstitial Pneumonitis - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage - Grade 5 (Vascular disorders) | 1 (1) | 0 (0)
Labial lesion - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain - labial - Grade 3 (General disorders) | 1 (1) | 0 (0)
Edema - Labia - Grade 3 (Vascular disorders) | 1 (1) | 0 (0)
Weakness - Lower extremity - Grade 3 (General disorders) | 0 (0) | 1 (1)
Left Ventricular Systolic Dysfunction - Grade 3 (Cardiac disorders) | 0 (0) | 1 (1)
Lung Infection - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
Meningitis - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
Mental Status Change - Grade 3 (Psychiatric disorders) | 0 (0) | 1 (1)
Mucositis - Grade 3 (Infections and infestations) | 1 (1) | 1 (1)
Multisystem organ failure - Grade 4 (General disorders) | 0 (0) | 1 (1)
Multisystem organ failure - Grade 5 (General disorders) | 1 (1) | 1 (1)
Pain - Abdominal - Grade 3 (General disorders) | 1 (1) | 0 (0)
Pain - Right lower quadrant - Grade 3 (General disorders) | 1 (1) | 0 (0)
Pleural Effusion - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis - Grade 3 (Infections and infestations) | 3 (3) | 4 (4)
Pneumonitis - Grade 4 (Infections and infestations) | 0 (0) | 1 (1)
Poor engraftment - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pulmonary Embolism - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Infiltrates - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Infiltrates - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulseless electrical activity - Grade 5 (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory Failure - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory Failure - Grade 5 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Seizure - Grade 3 (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis - Grade 4 (Infections and infestations) | 2 (2) | 1 (1)
Sepsis - Grade 5 (Infections and infestations) | 0 (0) | 1 (1)
Slow engraftment - Grade 3 (Immune system disorders) | 0 (0) | 1 (1)
Stroke - Grade 2 (Nervous system disorders) | 0 (0) | 1 (1)
Syncope - Grade 3 (Nervous system disorders) | 1 (1) | 4 (4)
Thrombocytopenia - Grade 4 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urinary Tract Infection - Grade 3 (Infections and infestations) | 0 (0) | 1 (1)
Fungal Infection - Grade 5 (Infections and infestations) | 0 (0) | 1 (1)
Blood and Lymphatic System Disorders - Other - Grade 5 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heart Failure - Grade 5 (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative HSCT (N=33) | Reduced Intensity HSCT (N=45)
Abdominal Distention - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Abdominal Distention - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Abnormal DLCO test - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abrasion - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acute Kidney Injury - Grade 1 (Renal and urinary disorders) | 5 (6) | 9 (10)
Acute Kidney Injury - Grade 2 (Renal and urinary disorders) | 3 (3) | 3 (3)
Acute Respiratory Acidosis - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adrenal adenoma - Grade 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Agitation - Grade 1 (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation - Grade 2 (Psychiatric disorders) | 0 (0) | 4 (4)
Agitation - Grade 4 (Psychiatric disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased - Grade 2 (Hepatobiliary disorders) | 2 (2) | 6 (6)
Alanine aminotransferase increased - Grade 2 (Hepatobiliary disorders) | 2 (2) | 0 (0)
Alanine phosphatase increased - Grade 1 (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic rhinitis - Grade 1 (Immune system disorders) | 0 (0) | 2 (2)
Alloimmunization - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Alopecia - Grade 1 (Immune system disorders) | 7 (7) | 5 (5)
Alopecia - Grade 2 (Immune system disorders) | 1 (1) | 0 (0)
Altered Mental State - Grade 1 (Psychiatric disorders) | 1 (1) | 0 (0)
Altered Taste - Grade 2 (General disorders) | 0 (0) | 2 (2)
Anal fistula - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anasarca - Grade 2 (General disorders) | 0 (0) | 1 (1)
Angina pectoris - Grade 1 (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris - Grade 2 (Cardiac disorders) | 1 (1) | 0 (0)
Anorexia - Grade 1 (Psychiatric disorders) | 1 (1) | 5 (5)
Anorexia - Grade 2 (Psychiatric disorders) | 6 (6) | 8 (8)
Anorexia - Grade 3 (Psychiatric disorders) | 5 (5) | 5 (5)
Anxiety - Grade 1 (Psychiatric disorders) | 9 (10) | 15 (18)
Anxiety - Grade 2 (Psychiatric disorders) | 15 (15) | 17 (18)
Aphthous ulcer - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aphthous ulcer - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arrhythmia - Grade 1 (Cardiac disorders) | 3 (3) | 2 (2)
Arrhythmia - Grade 2 (Cardiac disorders) | 3 (3) | 2 (2)
Arthraglia - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (10)
Arthraglia - Grade 2 (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (9)
Arthraglia - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ascites - Grade 1 (Vascular disorders) | 1 (1) | 1 (1)
Ascites - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Aseptic Meningitis - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased - Grade 1 (Hepatobiliary disorders) | 3 (3) | 6 (6)
Aspiration - Grade 2 (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Asthenia - Grade 2 (General disorders) | 1 (1) | 0 (0)
Asthma - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Atelectasis - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial Fibrillation - Grade 2 (Cardiac disorders) | 3 (4) | 4 (6)
Atrial tachycardia - Grade 2 (Cardiac disorders) | 0 (0) | 1 (1)
Awakening to Urinate - Grade 1 (Renal and urinary disorders) | 7 (7) | 9 (9)
Bacteremia - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia - Grade 3 (Infections and infestations) | 4 (4) | 5 (5)
Balance Problems - Grade 1 (Nervous system disorders) | 3 (3) | 3 (3)
Barodontalgia - Grade 1 (General disorders) | 0 (0) | 1 (1)
Behavioral Issues - Grade 2 (Psychiatric disorders) | 0 (0) | 1 (1)
BK Viremia - Grade 1 (Infections and infestations) | 1 (1) | 1 (1)
BK Viremia - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
BK Viremia - Grade 3 (Infections and infestations) | 0 (0) | 1 (1)
BK Virus Cystitis - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
Bleeding - Grade 1 (General disorders) | 1 (1) | 1 (1)
Blister - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Bloating - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating - Grade 2 (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blurred Vision - Grade 1 (Eye disorders) | 4 (4) | 7 (8)
Blurred Vision - Grade 2 (Eye disorders) | 2 (2) | 0 (0)
Bradycardia - Grade 1 (Cardiac disorders) | 4 (5) | 2 (2)
Bradycardia - Grade 2 (Cardiac disorders) | 2 (2) | 3 (3)
Bronchitis - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bruising - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Burning Ears - Grade 1 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Burning Palms - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Candidemia - Grade 3 (Infections and infestations) | 0 (0) | 1 (1)
Cardiac - Abnormal T wave - Grade 1 (Cardiac disorders) | 1 (1) | 0 (0)
Celiac artery stenosis - Grade 1 (Vascular disorders) | 1 (1) | 0 (0)
Cellulitis - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Change in Mental Status - Grade 2 (Psychiatric disorders) | 2 (2) | 1 (1)
Change in Vision - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Charcot Foot - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Charcot Joint - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chipped tooth - Grade 1 (General disorders) | 0 (0) | 1 (1)
Cholelithiasis - Grade 1 (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic Kidney Disease - Grade 1 (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Renal Failure - Grade 1 (Renal and urinary disorders) | 1 (1) | 0 (0)
Clostridium Difficile Infection - Grade 1 (Infections and infestations) | 1 (1) | 3 (3)
Clostridium Difficile Infection - Grade 2 (Infections and infestations) | 3 (3) | 2 (3)
CMV Reactivation - Grade 1 (Infections and infestations) | 3 (3) | 1 (1)
CMV Reactivation - Grade 2 (Infections and infestations) | 5 (6) | 3 (3)
CMV Viremia - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
CMV Viremia - Grade 2 (Infections and infestations) | 1 (1) | 2 (2)
CMV Viremia - Grade 3 (Infections and infestations) | 0 (0) | 3 (3)
Colitis - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Concentration impairment - Grade 1 (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion - Grade 1 (Psychiatric disorders) | 4 (4) | 8 (11)
Confusion - Grade 2 (Psychiatric disorders) | 6 (6) | 4 (5)
Congestion - Grade 1 (Immune system disorders) | 7 (7) | 1 (1)
Congestion - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Conjunctival Hemorrhage - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Conjunctival Hemorrhage - Grade 2 (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis - Grade 2 (Eye disorders) | 1 (1) | 2 (2)
Constipation - Grade 1 (Gastrointestinal disorders) | 13 (16) | 23 (39)
Constipation - Grade 2 (Gastrointestinal disorders) | 2 (3) | 2 (2)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cramping - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cystitis - Grade 2 (Renal and urinary disorders) | 0 (0) | 2 (2)
Cystitis - Grade 3 (Renal and urinary disorders) | 1 (1) | 0 (0)
Cytokine Release Syndrome - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Deconditioning - Grade 1 (General disorders) | 1 (1) | 0 (0)
Deconditioning - Grade 2 (General disorders) | 0 (0) | 1 (1)
Deconditioning - Grade 3 (General disorders) | 0 (0) | 1 (1)
decreased concentration - Grade 1 (Psychiatric disorders) | 1 (1) | 1 (1)
Decreased Ejection Fraction - Grade 2 (Cardiac disorders) | 0 (0) | 2 (2)
Decreased Hearing - L ear - Grade 2 (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Decreased urine retention - Grade 2 (Renal and urinary disorders) | 0 (0) | 1 (1)
Decreased Visual Focus - Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Decreased/coarse Breath Sounds - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dehydration - Grade 1 (General disorders) | 1 (1) | 0 (0)
Dehydration - Grade 2 (General disorders) | 5 (5) | 7 (7)
Delirium - Grade 2 (Psychiatric disorders) | 0 (0) | 1 (1)
Depression - Grade 1 (Psychiatric disorders) | 8 (8) | 8 (8)
Depression - Grade 2 (Psychiatric disorders) | 7 (7) | 10 (10)
Detrusor contraction - Grade 2 (Renal and urinary disorders) | 1 (1) | 1 (1)
Diabetes - Type 2 - Grade 1 (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diaphoresis - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Diarrhea - Grade 1 (Gastrointestinal disorders) | 16 (19) | 15 (19)
Diarrhea - Grade 2 (General disorders) | 9 (14) | 18 (23)
Diarrhea - Grade 3 (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diplopia - Grade 2 (Eye disorders) | 0 (0) | 1 (1)
Distressed - Grade 2 (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness - Grade 1 (Ear and labyrinth disorders) | 6 (8) | 12 (15)
Dizziness - Grade 2 (Ear and labyrinth disorders) | 4 (5) | 9 (12)
Dry Eye - Grade 1 (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Dry Eyes - Grade 2 (Eye disorders) | 1 (1) | 1 (1)
Dry Lips - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry Nasal passages - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry Skin - Grade 1 (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5)
Dry Skin - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DVT - Grade 2 (Vascular disorders) | 2 (2) | 2 (2)
DVT - Pericatheter Thrombus - Grade 2 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dysgeusia - Grade 1 (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dysgeusia - Grade 2 (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia - Grade 1 (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dyspepsia - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia - Grade 1 (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dysphagia - Grade 2 (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dyspnea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 13 (16)
Dyspnea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Dyspnea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea on Exertion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Dyspnea on Exertion - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dysuria - Grade 1 (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria - Grade 2 (Renal and urinary disorders) | 0 (0) | 7 (7)
Ear Fullness - grade 1 (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear Wax - Grade 1 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eczema - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Edema - Grade 1 (Vascular disorders) | 6 (6) | 2 (2)
Edema - Grade 2 (Vascular disorders) | 2 (2) | 1 (1)
Edema - Ankle - Grade 1 (Vascular disorders) | 2 (2) | 1 (1)
Edema - Arm - Grade 1 (Vascular disorders) | 2 (3) | 1 (1)
Edema - Arytenoid - Grade 2 (Vascular disorders) | 1 (1) | 0 (0)
Edema - Elbow - Grade 2 (Vascular disorders) | 1 (1) | 0 (0)
Edema - Extremities - Grade 1 (Vascular disorders) | 6 (7) | 23 (23)
Edema - Extremities - Grade 2 (Vascular disorders) | 1 (1) | 4 (4)
Edema - Eye - Grade 1 (Vascular disorders) | 0 (0) | 2 (2)
Edema - Eye Lid - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Edema - Face - Grade 1 (Vascular disorders) | 2 (2) | 3 (3)
Edema - Foot - Grade 1 (Vascular disorders) | 0 (0) | 1 (1)
Edema - Genital - Grade 2 (Vascular disorders) | 2 (2) | 0 (0)
Edema - Groin - Grade 1 (Vascular disorders) | 0 (0) | 2 (2)
Edema - Hand - Grade 1 (Vascular disorders) | 3 (3) | 1 (1)
Edema - Jaw - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Edema - Knees - Grade 1 (Vascular disorders) | 0 (0) | 1 (1)
Edema - Neck - Grade 1 (Vascular disorders) | 0 (0) | 2 (2)
Edema - Neck - Grade 2 (Vascular disorders) | 1 (1) | 0 (0)
Edema - Periorbial - Grade 1 (Vascular disorders) | 0 (0) | 2 (2)
Ejection Fraction Decreased - Grade 2 (Cardiac disorders) | 1 (1) | 1 (1)
Electrolyte Imbalance - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Electrolyte Imbalance - Grade 2 (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Electrolyte Imbalance - Grade 3 (Blood and lymphatic system disorders) | 2 (2) | 7 (7)
Elevated alkaline phosphatase - Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated ferritin - Grade 1 (Hepatobiliary disorders) | 0 (0) | 2 (2)
Elevated ferritin - Grade 2 (Hepatobiliary disorders) | 1 (1) | 0 (0)
Elevated Liver Function Tests - Grade 1 (Hepatobiliary disorders) | 1 (1) | 4 (4)
Elevated Liver Function Tests - Grade 2 (Hepatobiliary disorders) | 1 (1) | 2 (2)
Elevated Liver Function Tests - Grade 3 (Hepatobiliary disorders) | 2 (2) | 0 (0)
Elevated Prostate Specific Antigen - Grade 1 (Renal and urinary disorders) | 0 (0) | 1 (1)
Elevated Thyroid Stimulating Hormone - Grade 1 (Endocrine disorders) | 0 (0) | 1 (1)
Emesis - Grade 1 (Gastrointestinal disorders) | 8 (13) | 14 (17)
Emesis - Grade 2 (Gastrointestinal disorders) | 0 (0) | 5 (5)
Enlarged prostate - Grade 1 (Renal and urinary disorders) | 0 (0) | 1 (1)
Epigastric Burning - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epiphora - Grade 1 (Eye disorders) | 4 (4) | 0 (0)
Epistaxis - Grade 1 (Vascular disorders) | 2 (2) | 7 (8)
Epistaxis - Grade 2 (Vascular disorders) | 1 (1) | 2 (2)
Epistaxis - Grade 3 (Vascular disorders) | 0 (0) | 1 (1)
Epstein-Barr virus (EBV) positive - Grade 1 (Infections and infestations) | 0 (0) | 1 (1)
Erectile Dysfunction - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Erythema - Grade 1 (Vascular disorders) | 4 (5) | 5 (7)
Erythema - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Erythema - Grade 3 (Vascular disorders) | 1 (1) | 0 (0)
Erythema Multiforme - Grade 1 (Vascular disorders) | 0 (0) | 1 (1)
Erythema Multiforme - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Erythroderma - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythroderma - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Esophagitis - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis - Grade 3 (Gastrointestinal disorders) | 4 (4) | 2 (2)
Eustachian tube dysfunction - Grade 1 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excoriation - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Excoriation - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eye Problems - Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Eye ptosis - Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Facial numbness - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Facial Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Fall - Grade 1 (General disorders) | 0 (0) | 1 (1)
Fall - Grade 2 (General disorders) | 0 (0) | 4 (5)
Fatigue - Grade 1 (General disorders) | 4 (4) | 4 (4)
Fatigue - Grade 2 (General disorders) | 18 (20) | 27 (27)
Fatigue - Grade 3 (General disorders) | 9 (9) | 13 (13)
Fever - Grade 1 (Immune system disorders) | 23 (47) | 40 (66)
Fever - Grade 2 (Immune system disorders) | 17 (22) | 9 (14)
Fever - Grade 3 (Immune system disorders) | 3 (3) | 8 (12)
Fibrinogen decreased - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Flatulence - Grade 1 (Gastrointestinal disorders) | 2 (3) | 5 (5)
Flatulence - Grade 2 (Gastrointestinal disorders) | 1 (1) | 1 (1)
Floaters - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Fluid Filled Blister - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fluid Overload - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fluid Overload - Grade 2 (Blood and lymphatic system disorders) | 8 (8) | 8 (9)
Flushing - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Folliculitis - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Foot Redness - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fracture - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fungal Rash - Grade 1 (Infections and infestations) | 0 (0) | 1 (1)
Gait disturbance - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Gait disturbance - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastritis - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastroesophageal reflux disease - Grade 1 (Gastrointestinal disorders) | 1 (1) | 1 (1)
gastroesophageal reflux disease - Grade 2 (Gastrointestinal disorders) | 7 (7) | 11 (11)
Gilbert's Syndrome - Grade 1 (Hepatobiliary disorders) | 1 (1) | 0 (0)
Glass opacity in the lung - Grade 2 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gout - Grade 2 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hallucinations - Grade 1 (Psychiatric disorders) | 3 (3) | 3 (3)
Hallucinations - Grade 2 (Psychiatric disorders) | 0 (0) | 1 (1)
Headache - Grade 1 (General disorders) | 8 (10) | 8 (11)
Headache - Grade 2 (General disorders) | 8 (9) | 11 (11)
Hearing Problems - Grade 1 (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Hearing Problems - Grade 2 (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Heart Failure - Grade 2 (Cardiac disorders) | 1 (1) | 0 (0)
Hematochezia - Grade 1 (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hematoma - Grade 1 (Vascular disorders) | 0 (0) | 1 (1)
Hematoma - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Hematuria - Grade 1 (Blood and lymphatic system disorders) | 2 (2) | 7 (8)
Hematuria - Grade 2 (Blood and lymphatic system disorders) | 1 (1) | 7 (7)
Hemochromatosis - Grade 1 (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hemochromatosis - Grade 2 (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hemochromatosis - Grade 3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoptysis - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hemoptysis - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage - Oral - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hemorrhage - Oral - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hemorrhage - Right Eye - Grade 1 (Eye disorders) | 2 (2) | 0 (0)
Hemorrhoids - Grade 1 (Vascular disorders) | 1 (1) | 5 (5)
Hemorrhoids - Grade 2 (Vascular disorders) | 2 (2) | 0 (0)
Hepatitis B - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Hernia - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HHV-6 DNAemia - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
HHV-6 Viremia - Grade 1 (Infections and infestations) | 2 (2) | 3 (3)
HHV-6 Viremia - Grade 2 (Infections and infestations) | 1 (1) | 2 (2)
HHV-6 Viremia - Grade 3 (Infections and infestations) | 2 (2) | 1 (1)
Hoarseness - Grade 1 (General disorders) | 2 (2) | 1 (1)
Hordeolum externum - Grade 2 (Eye disorders) | 1 (2) | 0 (0)
Hot flashes - Grade 1 (General disorders) | 1 (1) | 0 (0)
hyperalkalinephosphatasemia - Grade 1 (Hepatobiliary disorders) | 1 (1) | 5 (5)
Hyperbilirubinemia - Grade 1 (Hepatobiliary disorders) | 8 (9) | 12 (13)
Hyperbilirubinemia - Grade 2 (Hepatobiliary disorders) | 5 (5) | 7 (7)
Hyperbilirubinemia - Grade 3 (Hepatobiliary disorders) | 1 (1) | 4 (4)
Hyperbilirubinemia - Grade 4 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperglycemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperhidrosis - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkalemia - Grade 1 (Renal and urinary disorders) | 1 (1) | 1 (1)
Hyperkalemia - Grade 2 (Renal and urinary disorders) | 1 (1) | 2 (2)
Hyperkalemia - Grade 3 (Renal and urinary disorders) | 1 (1) | 2 (2)
Hyperlipidemia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Hyperlipidemia - Grade 2 (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hypernatremia - Grade 1 (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypernatremia - Grade 2 (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypernatremia - Grade 3 (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertension - Grade 1 (Vascular disorders) | 12 (13) | 9 (9)
Hypertension - Grade 2 (Vascular disorders) | 13 (15) | 22 (23)
hypervolemia - grade 1 (Vascular disorders) | 1 (1) | 2 (2)
hypervolemia - Grade 2 (Vascular disorders) | 4 (4) | 5 (5)
hypoesthesia - right upper quadrant - Grade 1 (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycemia - Grade 1 (Endocrine disorders) | 2 (2) | 1 (1)
hypogonadism - Grade 2 (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypokalemia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypokalemia - Grade 3 (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Hypomagnesemia - Grade 1 (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypomagnesemia - Grade 2 (Renal and urinary disorders) | 2 (2) | 1 (1)
Hypomagnesemia - Grade 3 (Renal and urinary disorders) | 0 (0) | 2 (2)
Hyponatremia - Grade 1 (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hyponatremia - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypophosphatemia - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypotension - Grade 1 (Cardiac disorders) | 4 (4) | 10 (11)
Hypotension - Grade 2 (Cardiac disorders) | 14 (17) | 21 (30)
Hypotension - Grade 3 (Cardiac disorders) | 1 (1) | 2 (2)
Hypothermia - Grade 2 (General disorders) | 2 (3) | 3 (3)
Hypothyroidism - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypoxia - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (9)
Hypoxia - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Immune thrombocytopenic purpura - Grade 2 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Impaired fasting glucose - Grade 2 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Impulsivity - Grade 1 (Psychiatric disorders) | 0 (0) | 1 (1)
Increased Acute Rheumatic Fever - Grade 2 (Cardiac disorders) | 0 (0) | 1 (1)
Increased Alkaline Phosphatase - Grade 1 (Hepatobiliary disorders) | 1 (1) | 1 (1)
Increased Creatinine - Grade 1 (Renal and urinary disorders) | 6 (6) | 6 (8)
Increased Creatinine - Grade 2 (Renal and urinary disorders) | 1 (1) | 2 (2)
Increased Ferritin - Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Increased Liver Function Tests - Grade 1 (Hepatobiliary disorders) | 1 (1) | 1 (1)
Increased Liver Function Tests - Grade 2 (Hepatobiliary disorders) | 2 (2) | 1 (1)
Increased Urination - Grade 1 (Renal and urinary disorders) | 0 (0) | 1 (1)
Indigestion - Grade 1 (Gastrointestinal disorders) | 1 (1) | 1 (1)
Indigestion - Grade 2 (Gastrointestinal disorders) | 3 (3) | 4 (4)
Infection and Infestations - Other - Grade 3 (Infections and infestations) | 2 (2) | 0 (0)
Infectious Diarrhea - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction - bradycardia - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Chest pain - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Chills - Grade 1 (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Infusion Related Reaction - Chest tightness - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Chills - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Infusion related reaction - dizziness - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction - eye floaters - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction - fatigue - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Fever - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Fever - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Infusion Related Reaction - Flushing - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Hives - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Hives - Grade 2 (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Infusion Related Reaction - Hives - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - HSCT - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Hypotension - Grade 1 (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Infusion Related Reaction - Hypotension - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Hypotension - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Itching - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - IVIG - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Nausea - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Infusion Related Reaction - Nausea - Grade 2 (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infusion Related Reaction - Nausea - Grade 4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Numbness - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Platelets - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - PLTs - Grade 2 (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Infusion Related Reaction - Pruritis - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Rash - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Rash - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Infusion Related Reaction - Rigors - Grade 1 (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infusion Related Reaction - Rigors - Grade 2 (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Infusion Related Reaction - SOB - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Tachycardia - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Tachycardia - Grade 2 (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Infusion Related Reaction - unspecified - Grade 1 (Injury, poisoning and procedural complications) | 3 (6) | 0 (0)
Infusion Related Reaction - unspecified - Grade 2 (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Infusion Related Reaction - unspecified - Grade 3 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Vomiting - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction - Vomiting - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inguinal hernia - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Insomnia - Grade 1 (Psychiatric disorders) | 20 (25) | 17 (18)
Insomnia - Grade 2 (Psychiatric disorders) | 0 (0) | 10 (12)
Intracranial Hemorrhage - Grade 2 (Vascular disorders) | 1 (1) | 0 (0)
Irritable - Grade 1 (Psychiatric disorders) | 1 (1) | 0 (0)
Irritable - Grade 2 (Psychiatric disorders) | 1 (1) | 1 (1)
Itching Throat - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Itchy Eyes - Grade 2 (Eye disorders) | 0 (0) | 1 (1)
Laceration - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lack of Taste - Grade 1 (General disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction - Grade 2 (Cardiac disorders) | 0 (0) | 1 (1)
Leg Cramps - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lesion - Rectum - Grade 1 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lesion - Penis - Grade 1 (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lethargy - Grade 1 (General disorders) | 0 (0) | 1 (1)
Lethargy - Grade 2 (General disorders) | 2 (2) | 3 (3)
Lethargy - Grade 3 (General disorders) | 0 (0) | 1 (1)
Lipoma - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Liver Cyst - Grade 1 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lung Infection - Grade 2 (Immune system disorders) | 2 (2) | 1 (1)
Lung nodule - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lymphocytosis - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Malaise - Grade 2 (General disorders) | 1 (1) | 1 (2)
Memory change - Grade 1 (Psychiatric disorders) | 2 (2) | 0 (0)
Menorrhagia - Grade 2 (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Metabolic Alkalosis - Grade 1 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Migraine - Grade 1 (General disorders) | 0 (0) | 1 (1)
Migraine - Grade 2 (General disorders) | 0 (0) | 1 (1)
Mitral valve disease - Grade 1 (Cardiac disorders) | 0 (0) | 1 (1)
Mobitz Type I - Grade 2 (Cardiac disorders) | 0 (0) | 1 (1)
Mole - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
monoclonal gammopathy of unknown significance - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mood Changes - Grade 1 (Psychiatric disorders) | 0 (0) | 1 (1)
Mouth - Thick Mucous Secretions - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Changes - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Mucositis - Grade 1 (Gastrointestinal disorders) | 1 (1) | 8 (9)
Mucositis - Grade 2 (Gastrointestinal disorders) | 6 (7) | 10 (11)
Mucositis - Grade 3 (Gastrointestinal disorders) | 23 (23) | 14 (14)
Murmur - Grade 1 (Cardiac disorders) | 2 (2) | 2 (2)
Myalgia - Grade 1 (General disorders) | 2 (2) | 1 (1)
Myalgia - Grade 2 (General disorders) | 1 (1) | 2 (2)
Nails Peeling - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nasal Congestion - Grade 1 (Immune system disorders) | 4 (4) | 1 (1)
Nasal Congestion - Grade 2 (Immune system disorders) | 1 (1) | 1 (1)
Nasal Discharge - Grade 1 (Immune system disorders) | 1 (1) | 0 (0)
Nasal Dryness - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea - Grade 1 (Gastrointestinal disorders) | 5 (5) | 4 (4)
Nausea - Grade 2 (Gastrointestinal disorders) | 10 (12) | 12 (12)
Nausea - Grade 3 (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neuralgia - Grade 2 (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy - Grade 1 (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy - Grade 2 (Nervous system disorders) | 1 (1) | 5 (5)
Nocturia - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Nocturia - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nonspecific skin eruption - grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Obesity - Grade 2 (General disorders) | 1 (1) | 1 (1)
Obesity - Grade 3 (General disorders) | 1 (1) | 2 (2)
Obesity - Grade 4 (General disorders) | 1 (1) | 0 (0)
Obstructive Sleep Apnea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Odynophagia - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oliguria - Grade 1 (Renal and urinary disorders) | 4 (4) | 0 (0)
Oliguria - Grade 2 (Renal and urinary disorders) | 11 (14) | 13 (15)
Orthostatic Hypotension - Grade 2 (Nervous system disorders) | 4 (4) | 3 (3)
Orthostatic Hypotension - Grade 3 (Nervous system disorders) | 0 (0) | 1 (1)
Oseomyelitis - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Osteopenia - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis - Grade 2 (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain - Abdominal - Grade 1 (General disorders) | 8 (11) | 12 (12)
Pain - Abdominal - Grade 2 (General disorders) | 12 (15) | 15 (20)
Pain - Arm - Grade 1 (General disorders) | 2 (2) | 1 (1)
Pain - Arm - Grade 2 (General disorders) | 1 (1) | 1 (1)
Pain - B/L Hips/thighs - Grade 1 (General disorders) | 0 (0) | 1 (1)
Pain - Back - Grade 1 (General disorders) | 8 (8) | 4 (6)
Pain - Back - Grade 2 (General disorders) | 4 (4) | 8 (8)
Pain - Back - Grade 3 (General disorders) | 0 (0) | 1 (1)
Pain - BM site - Grade 2 (General disorders) | 1 (1) | 0 (0)
Pain - Bone - Grade 1 (General disorders) | 1 (1) | 1 (1)
Pain - Bone - Grade 2 (General disorders) | 2 (2) | 1 (1)
Pain - Buttocks - Grade 2 (General disorders) | 0 (0) | 1 (1)
Pain - Calf - Grade 1 (General disorders) | 0 (0) | 1 (1)
Pain - Calf - Grade 2 (General disorders) | 0 (0) | 1 (1)
Pain - Catheter site - Grade 1 (General disorders) | 0 (0) | 2 (2)
Pain - Chest - Grade 1 (General disorders) | 8 (11) | 4 (6)
Pain - Chest - Grade 2 (General disorders) | 4 (4) | 4 (4)
Pain - Ear - Grade 1 (General disorders) | 0 (0) | 2 (2)
Pain - Elbow - Grade 1 (General disorders) | 1 (1) | 1 (1)
Pain - Epigastric - Grade 1 (General disorders) | 1 (1) | 1 (1)
Pain - Epigastric - Grade 2 (General disorders) | 1 (1) | 0 (0)
Pain - Extremities - Grade 1 (General disorders) | 4 (4) | 2 (2)
Pain - Extremities - Grade 2 (General disorders) | 3 (3) | 1 (1)
Pain - Eye - Grade 1 (General disorders) | 3 (3) | 1 (1)
Pain - Face - Grade 1 (General disorders) | 0 (0) | 3 (3)
Pain - Face - Grade 2 (General disorders) | 0 (0) | 1 (1)
Pain - Feet - Grade 1 (General disorders) | 1 (2) | 0 (0)
Pain - Flank - Grade 1 (General disorders) | 2 (2) | 1 (1)
Pain - Flank - Grade 2 (General disorders) | 1 (1) | 0 (0)
Pain - Foley Insertion Site - Grade 1 (General disorders) | 0 (0) | 1 (1)
Pain - Foot - Grade 2 (General disorders) | 2 (2) | 0 (0)
Pain - Groin - Grade 1 (General disorders) | 1 (1) | 0 (0)
Pain - Hand - Grade 1 (General disorders) | 1 (1) | 1 (1)
Pain - Hand - Grade 2 (General disorders) | 1 (1) | 1 (1)
Pain - Heel - Grade 1 (General disorders) | 1 (1) | 0 (0)
Pain - Hemorrhoids - Grade 2 (General disorders) | 1 (1) | 0 (0)
Pain - Hip - Grade 1 (General disorders) | 1 (1) | 0 (0)
Pain - Hip - Grade 2 (General disorders) | 1 (1) | 2 (2)
Pain - Jaw - Grade 1 (General disorders) | 0 (0) | 1 (1)
Pain - Jaw - Grade 2 (General disorders) | 3 (3) | 1 (1)
Pain - Knee - Grade 1 (General disorders) | 1 (1) | 1 (1)
Pain - Knee - Grade 2 (General disorders) | 2 (2) | 1 (1)
Pain - Left Upper Quadrant - Grade 2 (General disorders) | 0 (0) | 1 (1)
Pain - Leg - Grade 2 (General disorders) | 1 (2) | 1 (1)
Pain - Muscle - Grade 1 (General disorders) | 1 (1) | 2 (2)
Pain - Muscle - Grade 2 (General disorders) | 2 (2) | 1 (1)
Pain - Neck - Grade 1 (General disorders) | 4 (4) | 2 (2)
Pain - Neck - Grade 2 (General disorders) | 3 (3) | 2 (3)
Pain - Neck - Grade 3 (General disorders) | 0 (0) | 1 (1)
Pain - Oral - Grade 1 (General disorders) | 0 (0) | 1 (1)
Pain - Oral - Grade 2 (General disorders) | 0 (0) | 1 (1)
Pain - Pelvic - Grade 1 (General disorders) | 2 (2) | 0 (0)
Pain - Penile - Grade 1 (General disorders) | 1 (1) | 0 (0)
Pain - Penile - Grade 2 (General disorders) | 2 (2) | 1 (1)
Pain - Penile - Grade 3 (General disorders) | 1 (1) | 0 (0)
Pain - PICC site - Grade 1 (General disorders) | 1 (2) | 0 (0)
Pain - PICC site - Grade 2 (General disorders) | 2 (3) | 0 (0)
Pain - rectal - Grade 1 (General disorders) | 3 (4) | 1 (1)
Pain - rectal - Grade 2 (General disorders) | 3 (3) | 0 (0)
Pain - Scrotal - Grade 2 (General disorders) | 1 (1) | 2 (2)
Pain - Shoulder - Grade 1 (General disorders) | 2 (2) | 1 (1)
Pain - Shoulder - Grade 2 (General disorders) | 2 (2) | 1 (1)
Pain - Shoulder - Grade 3 (General disorders) | 0 (0) | 1 (1)
Pain - Sinus - Grade 1 (General disorders) | 1 (1) | 1 (1)
Pain - Skin - Grade 1 (General disorders) | 1 (1) | 0 (0)
Pain - Teeth - Grade 1 (General disorders) | 1 (1) | 0 (0)
Pain - Throat - Grade 1 (General disorders) | 1 (1) | 0 (0)
Pain - Throat - Grade 2 (General disorders) | 0 (0) | 1 (1)
Pain - Toe - Grade 1 (General disorders) | 1 (1) | 0 (0)
Pain - Urinary - Grade 1 (General disorders) | 1 (1) | 3 (4)
Pain - Wrist - Grade 1 (General disorders) | 0 (0) | 1 (1)
Pallor - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Parainfluenza 3 - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Paresthesia - Grade 1 (Nervous system disorders) | 6 (6) | 9 (9)
Paresthesia - Grade 2 (Nervous system disorders) | 1 (1) | 2 (2)
Paresthesia - Foot - Grade 1 (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesia - Mouth - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Parotitis - Grade 1 (Injury, poisoning and procedural complications) | 5 (6) | 0 (0)
Parotitis - Grade 2 (Vascular disorders) | 1 (1) | 0 (0)
Penile spasms - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pericardial Effusion - Grade 1 (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial Effusion - Grade 2 (Cardiac disorders) | 4 (4) | 2 (2)
Pericatheter Thrombus - Grade 2 (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Periorbital Redness - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Peripheral Motor Neuropathy - Grade 1 (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral Motor Neuropathy - Grade 2 (Nervous system disorders) | 2 (2) | 1 (1)
Perirectal Bleed - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Perirectal Irritation - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Perorbital Bruise - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pleural Effusion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleural Effusion - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural Effusion - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Hemorrhage - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pollakiuria - Grade 1 (Renal and urinary disorders) | 4 (5) | 8 (10)
Pollakiuria - Grade 2 (Renal and urinary disorders) | 2 (2) | 3 (3)
Poor Urine Output - Grade 1 (Renal and urinary disorders) | 1 (1) | 0 (0)
Postnasal drip - Grade 1 (Immune system disorders) | 2 (2) | 0 (0)
Pressure injury - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
presyncope - Grade 1 (Ear and labyrinth disorders) | 0 (0) | 3 (5)
presyncope - Grade 2 (Ear and labyrinth disorders) | 0 (0) | 4 (4)
Pruritus - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2) | 10 (12)
Pruritus - Grade 2 (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (6)
Ptysis - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary Edema - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Edema - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Hypertension - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Hypertension - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Infiltrates - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Infiltrates - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary nodules - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Premature Ventricular Contractions - Grade 1 (Cardiac disorders) | 0 (0) | 1 (1)
Pyschosis - Grade 2 (Psychiatric disorders) | 0 (0) | 1 (1)
Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 9 (10) | 29 (31)
Rash - Grade 2 (Skin and subcutaneous tissue disorders) | 17 (23) | 17 (20)
Rash - Grade 3 (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (5)
Rectal Itching - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rectal Mucositis - Grade 3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal insufficiency - Grade 1 (Renal and urinary disorders) | 1 (1) | 1 (1)
Rhinorrhea - Grade 1 (Immune system disorders) | 2 (2) | 0 (0)
Rhinorrhea - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Rhonchi - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rigors - Grade 1 (Nervous system disorders) | 11 (14) | 14 (17)
Rigors - Grade 2 (Nervous system disorders) | 0 (0) | 5 (5)
RSV B - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Sanguineous Drainage - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scabs - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scar - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Scattered skin tears - Grade 2 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scrotal Irritation - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seasonal Allergies - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Seizure - Grade 2 (Nervous system disorders) | 2 (2) | 0 (0)
Sensory Neuropathy - Grade 2 (Nervous system disorders) | 1 (1) | 0 (0)
Sexual Problems - Grade 1 (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Sibilant Rhonchus - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Singultus - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Singultus - Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Sinus Brachycardia - Grade 1 (Cardiac disorders) | 0 (0) | 4 (4)
Sinus Bradycardia - Grade 2 (Cardiac disorders) | 0 (0) | 2 (2)
Sinus Congestion - Grade 1 (Immune system disorders) | 0 (0) | 2 (2)
Sinus Congestion - Grade 2 (Immune system disorders) | 0 (0) | 2 (2)
Sinus Headache - Grade 1 (Immune system disorders) | 0 (0) | 1 (1)
Sinus Pressure - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Sinus Tachycardia - Grade 1 (Cardiac disorders) | 9 (15) | 9 (14)
Sinusitis - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis - Grade 2 (Infections and infestations) | 1 (1) | 1 (2)
Skin - Peeling - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discoloration - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hypopigmentation - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
skin induration - Grade 1 (Immune system disorders) | 1 (1) | 0 (0)
Skin infection - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Skin irritation - Grade 2 (Immune system disorders) | 1 (1) | 0 (0)
Skin irritation - Scrotum - Grade 1 (Immune system disorders) | 0 (0) | 1 (1)
Skin Lump - Grade 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin Nodules- Grade 1 (Immune system disorders) | 1 (1) | 0 (0)
Skin Nodules - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Skin Peeling - Grade 1 (Immune system disorders) | 1 (1) | 0 (0)
Skin Peeling - Grade 2 (Immune system disorders) | 0 (0) | 1 (1)
Skin Rash - GVHD - Grade 3 (Immune system disorders) | 1 (1) | 0 (0)
Skin tears - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin tightness - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sleep Apnea - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small Bowel Obstruction - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sneezing - Grade 1 (Immune system disorders) | 1 (1) | 0 (0)
Somnolence - Grade 1 (General disorders) | 1 (1) | 0 (0)
Sore Throat - Grade 1 (General disorders) | 3 (3) | 3 (3)
Sore Throat - Grade 2 (General disorders) | 0 (0) | 2 (2)
Speech change - Grade 1 (General disorders) | 2 (2) | 0 (0)
Subconjuctival hemorrhage - Grade 1 (Vascular disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia - Grade 1 (Cardiac disorders) | 0 (0) | 1 (1)
Sweating - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope - Grade 3 (Vascular disorders) | 0 (0) | 1 (1)
Syphilis - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Tachycardia - Grade 1 (Cardiac disorders) | 13 (14) | 15 (21)
Tachycardia - Grade 2 (Cardiac disorders) | 4 (4) | 3 (3)
Tachypnea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Tachypnea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tender Mass - RUE - Grade 1 (General disorders) | 1 (1) | 0 (0)
Tenderness - skin - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thromboembolic event - Grade 2 (Vascular disorders) | 2 (2) | 2 (2)
Thrush - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Thrush - Grade 2 (Infections and infestations) | 3 (3) | 3 (3)
Thyroid Nodule - Grade 1 (Endocrine disorders) | 0 (0) | 1 (1)
Transaminitis - Grade 2 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Tremor - Grade 1 (Nervous system disorders) | 5 (5) | 10 (11)
Tremor - Grade 2 (Nervous system disorders) | 1 (1) | 1 (1)
Tremor - Grade 3 (Nervous system disorders) | 1 (1) | 0 (0)
Tricuspid valve disease - Grade 1 (Cardiac disorders) | 1 (1) | 0 (0)
Tussis - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 11 (12)
Tussis - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Unsteadiness - Grade 1 (General disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection - Grade 1 (Infections and infestations) | 2 (2) | 0 (0)
Upper Respiratory Infection - Grade 2 (Infections and infestations) | 1 (1) | 1 (1)
Urethra irritation - Grade 1 (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency - Grade 1 (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence - Grade 1 (Renal and urinary disorders) | 3 (4) | 2 (2)
Urinary Incontinence - Grade 2 (Renal and urinary disorders) | 4 (4) | 5 (5)
Urinary Retention - Grade 1 (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary Retention - Grade 2 (Renal and urinary disorders) | 3 (3) | 4 (4)
Urinary Tract Infection - Grade 2 (Infections and infestations) | 3 (3) | 6 (6)
Urinary Tract Infection - Grade 3 (Infections and infestations) | 0 (0) | 1 (1)
Urinary Urgency - Grade 1 (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary Urgency - Grade 2 (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine Leiomyoma - Grade 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vaginal bleeding - Grade 1 (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Itching - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Venous stasis dermatitis - Grade 1 (Vascular disorders) | 1 (1) | 0 (0)
Vertigo - Grade 2 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Visual Hallucinations - Grade 1 (Psychiatric disorders) | 1 (1) | 2 (2)
Vitamin D deficiency - Grade 1 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency - Grade 2 (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Vivid Dreams - Grade 1 (Psychiatric disorders) | 5 (5) | 2 (2)
Vivid Dreams - Grade 2 (Psychiatric disorders) | 0 (0) | 1 (1)
Weakness - Lower extremity - Grade 1 (General disorders) | 4 (4) | 2 (2)
Weakness - Lower extremity - Grade 2 (General disorders) | 1 (1) | 1 (1)
Weakness - Right Side - Face - Grade 1 (General disorders) | 0 (0) | 1 (1)
Weight Loss - Grade 1 (General disorders) | 2 (2) | 3 (3)
Weight Loss - Grade 2 (General disorders) | 1 (1) | 2 (2)
Wound - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound - Back - Grade 1 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound - Buttocks - Grade 1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound - Elbow - Grade 1 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound - Sacrum - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound Bleeding - Grade 2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound - Skin - Grade 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Xerostomia - Grade 1 (Endocrine disorders) | 9 (11) | 5 (5)
Xerostomia - Grade 2 (Endocrine disorders) | 5 (5) | 0 (0)
Xerostomia - Grade 3 (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT01349101/Prot_SAP_000.pdf